CLINICAL TRIAL: NCT05570097
Title: Cryoanalgesia in Combination With the Novel Prehabilitation Program Back on Feet Are the Essential Parts of Enhanced Recovery Protocol in the Minimal Invasive Modyfied Nuss Procedure of Children With Funnel Chest Deformation.
Brief Title: Cryoanalgesia to Prevent Acute and Chronic Pain Following Nuss Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Principal Investigator, Sławomir Zacha, Principal Investigator, Pomeranian Medical University Szczecin
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PomeranianMedicalUniveristy
Record Dates: First submitted 2022-09-29; First posted 2022-10-06 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Funnel Chest; Excavatum, Pectus
Keywords: nuss procedure; ERAS; cryolesia; cryoanalgesia
MeSH Terms: conditions — Funnel Chest

STUDY DESIGN:
Intervention Model Description: Before - after study:
  First: control group as a standard treatment in Poland, review, then:
  interventional group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "the before" group (No Intervention): Control group as a standard therapy in Poland (regional analgesia: intrapleural or bilateral erector spine plane block added to multimodal analgesia).
- "the after" group (Experimental): During modyfied Nuss thoracoscopy the intraoperative Cryolesia of at least 5 intercostal nerves added to regional analgesia: bilateral erector spine plane block and multimodal therapy.
  Interventions: Device: intercostal nerves cryoanalgesia

INTERVENTIONS:
Device: intercostal nerves cryoanalgesia — Intraoperative Cryolesia of at least 5 intercostal nerves added to regional analgesia: bilateral erector spine plane block and multimodal therapy.
  Arms: "the after" group

SUMMARY:
This Study study compared standard therapy (multimodal and regional analgesia) versus a novel approach (Cryoanalgesia combined with bilateral erector spine plane block and multimodal analgesia) in subjects undergoing minimal invasive modyfied Nuss procedure (thoracoscopy).

DETAILED DESCRIPTION:
Funnel chest deformation is a great challenge for therapeutic teams due to severe pain in the postoperative period as well as chronic pain. The use of many analgesic drugs, including opioids, is associated with adverse side effects, difficulties with rehabilitation, an increased risk of complications, prolonged hospitalisation, and the cost of the procedure. Cryoanalgesia as a part of multimodal analgesia along with the education and prehabilitation of the patient according to the novel original educational - training application 'Back on Feet' as well as the interdisciplinary care in accordance with the enhanced recovery after surgery (ERAS) protocol, which has a real impact on the optimisation of perioperative care.

This Before - After Study is a single institution pilot study designed to compare standard therapy (control group: regional analgesia: intrapleural or bilateral erector spine plane block) versus a novel approach (interventional group: Cryoanalgesia combined with bilateral single shot erector spine plane block) to address the need for better management of acute and long-term pain in the pediatric population diagnosed with funnel-chest and treated using the modyfied Nuss method.

First group received a standard care according to Polish guidelines. The data of control group analysed and the interdisciplinary team work protocol will be introduced to the interventional group. The interventional group was prepared according to prehabilitation with the 'Back on feet' application and perioperative ERAS protocols. The patients of interventional group received intraoperative cryoanalgesia using the Cryo-S Painless device (Metrum - Cryoflex Polska Limited) as an additional procedure to multimodal analgesia. This is the first time that the cryoanalgesia procedure was performed in children in Poland.

The aims of the study were the assessment the effectiveness of cryoanalgesia as a method of acute and long-term pain control, safety of the method and the impact of preoperative preparation according to the 'Back on Feet' program introduced as a part of ERAS protocol.

Specific Aim 1: To determine if, compared with current analgesia, the addition of cryoanalgesia decreases the incidence and severity of post-surgical pain.

Hypothesis 1a (primary): The severity of surgically-related pain was significantly decreased from postoperative day 2 with the addition of cryoanalgesia as compared with patients receiving solely standard-of-care treatment.

Hypothesis 1b: The incidence and severity of chronic pain was significantly decreased 3 months following surgery with the addition of cryoanalgesia as compared with patients receiving solely standard-of-care treatment.

Specific Aim 2: To determine if, compared with current analgesia, the addition of cryoanalgesia improves postoperative functioning.

Hypothesis 2a: Following modyfied Nuss procedure the range of motion and independence was significantly increased in the 2 postoperative day following operation with the addition of cryoanalgesia as compared with patients receiving solely standard-of-care treatment.

The results were compared in terms of demographics, pain levels, side effects of the pain relief medications in the postoperative period, quality and length of rehabilitation, patient satisfaction using the Quality of Life by modyfied Nuss questionnaire, and the total costs of hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing pectus excavatum repair with modyfied minimal invasive thoracoscopic NUSS technique
* aged 10 years or above 10
* informed consent signed for cryoanalgesia

Exclusion Criteria:

* Age of 9 years or below
* Refuse to receive cryoanalgesia or regional analgesia as primary pain relief
* Any contraindication to cryoanalgesia
* Difficult follow-up for geographical reasons and/or impossibility by the patient to understand how to perform self-measurements

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-09-28 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-12-10 (Actual)

PRIMARY OUTCOMES:
The worse pain occurence during first 24 hours after operation | up to 24 hours after operation
  Numeric pain score. Range from 0 to 10.

SECONDARY OUTCOMES:
Analgesic consumption post operation | Postoperative days 0, 1, 2, 3, 4, 5,6, as well as months 1 and 3
  Total analgesic (including opioids) consumption for previous 24 hours
Thoracic hypo-aesthesia occurence | up to 24 hours after operation
  Cold test assessment (Yes/No)
Assessment of sleeping quality | Postoperative days 1, 2, 3, 4, 5 ,6
  Collect difficulties of sleeping due to pain? (binary answer: yes or no; not based on a scale or instrument)
Postoperative nausea and vomiting (PONV) occurence | Postoperative days 1, 2, 3, 4, 5 ,6
  binary answer: yes or no; not based on a scale or instrument
Residual wound or chest pain occurence | Postoperative months 1, 3
  The chest or wound chronic pain occurrences
Total narcotic use post-operation | 0-6 postoperative days
  Total dose and number of days of opioids used during hospitalization
Cost Analysis | estimated 1 week
  total costs of hospitalization
Duration of hospitalization | estimated 1 week
  the length of the time (in days) spent in the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Jowita Biernawska, MD PhD, Study Director — Pomeranian Medical Universitet Szczecin
Locations (1):
- Pomeranian Medical University, Szczecin, Poland

IPD SHARING:
Plan to Share IPD: Yes
We invite others researchers to collaboration as multicenter study.
Supporting Information: Study Protocol
Time Frame: up to 12 months from the beginning of the study
Access Criteria: by contact to Principal Investigator

REFERENCES:
- [Result] Graves CE, Moyer J, Zobel MJ, Mora R, Smith D, O'Day M, Padilla BE. Intraoperative intercostal nerve cryoablation During the Nuss procedure reduces length of stay and opioid requirement: A randomized clinical trial. J Pediatr Surg. 2019 Nov;54(11):2250-2256. doi: 10.1016/j.jpedsurg.2019.02.057. Epub 2019 Mar 17. PMID 30935731